CLINICAL TRIAL: NCT04385303
Title: A 28-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate a Single Injection of SM04690 Injected in the Target Knee Joint of Moderately to Severely Symptomatic Osteoarthritis Subjects
Brief Title: Patient-Reported Outcomes in Evaluating Lorecivivint (SM04690) for Moderate to Severe Knee Osteoarthritis (STRIDES-1)
Acronym: STRIDES-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SM04690-OA-10
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: SM04690; Wnt pathway inhibitor; osteoarthritis; Samumed; lorecivivint
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — lorecivivint

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vehicle (Active Comparator): Healthcare professional-administered intra-articular injection; performed on Day 1.
  Interventions: Drug: Placebo
- Lorecivivint (Experimental): Healthcare professional-administered intra-articular injection; performed on Day 1.
  Interventions: Drug: Lorecivivint

INTERVENTIONS:
Drug: Lorecivivint — One intra-articular injection of 0.07 mg lorecivivint in 2 mL vehicle
  Other Names: SM04690
  Arms: Lorecivivint
Drug: Placebo — One intra-articular injection of 0 mg lorecivivint in 2 mL vehicle
  Other Names: Vehicle
  Arms: Vehicle

SUMMARY:
This phase 3 study is a multicenter, randomized, double-blind, placebo-controlled study of lorecivivint injected intraarticularly (IA) into the target knee (most painful) joint of moderately to severely symptomatic osteoarthritis (OA) subjects at a single dose of 0.07 mg lorecivivint per 2 mL injection. This study will utilize patient reported outcomes (PROs) to evaluate the safety and efficacy of lorecivivint.

DETAILED DESCRIPTION:
SM04690-OA-10 was a phase 3, 28-week multicenter, randomized, double-blind, placebo-controlled, parallel group study investigating the safety, tolerability and efficacy of lorecivivint 0.07 mg (compared with placebo) injected into the target knee joint of moderately to severely symptomatic knee OA subjects.

Patient-reported outcomes included Pain Numeric Rating Scale (NRS) [0-10], Western Ontario and McMaster Universities Arthritis Index (WOMAC), and Patient Global Assessment (PGA) of knee osteoarthritis.

The primary efficacy endpoint was change from baseline in target knee Pain NRS at Week 12. Secondary endpoints included change at Week 12 in WOMAC Function and PGA.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females between 40 and 80 years of age, inclusive, in general good health apart from their knee OA
* Ambulatory (single assistive devices such as canes allowed if needed less than 50% of the time, subjects requiring a walker are excluded)
* Diagnosis of femorotibial OA in the target knee by standard American College of Rheumatology (ACR) criteria at the Screening Visit (clinical AND radiographic criteria); OA of the knee is not to be secondary to any rheumatologic conditions (e.g., rheumatoid arthritis)
* Radiographic disease Stage 2 or 3 in target knee within 24 weeks of the Screening Visit according to the Kellgren-Lawrence (KL) grading of knee OA as assessed by independent central readers
* Qualifying mean score on the 24-h average pain score (0-10 numeric rating scale)
* Pain compatible with OA of the knee(s) for at least 26 weeks prior to the Screening Visit
* Primary source of pain throughout the body is due to OA in the target knee
* Body mass index (BMI) ≤ 35 kg/m2 at the Screening Visit
* Negative drug test for amphetamine, buprenorphine, cocaine, methadone, opiates, phencyclidine (PCP), propoxyphene, barbiturates, benzodiazepine, methaqualone, and tricyclic antidepressants, unless any of these drugs are allowed per protocol and prescribed by a physician to treat a specific condition

Key Exclusion Criteria:

* Pregnant women, breastfeeding women, and women who are not post-menopausal (defined as 12 months with no menses without an alternative medical cause) or permanently surgically sterile (includes hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) who have a positive or indeterminate pregnancy test result at the Screening Visit or Day 1
* Significant malalignment of anatomical axis (medial angle formed by the femur and tibia) of the target knee (varus > 10°, valgus > 10°) by radiograph within 24 weeks of the Screening Visit as assessed by independent central readers
* Partial or complete joint replacement in either knee
* Currently requires use of a lower extremity prosthesis, and/or a structural knee brace (i.e., a knee brace that contains hardware)
* Any surgery (e.g., arthroscopy) in either knee within 26 weeks prior to Day 1
* Intra-articular (IA) injection into the target knee with a therapeutic aim including, but not limited to hyaluronic acid, platelet-rich plasma (PRP), and stem cell therapies within 26 weeks prior to Day 1; or IA glucocorticoids within 12 weeks prior to Day 1 allowed
* Previous treatment with lorecivivint (SM04690)
* Subjects who have previously failed screening on this protocol and fail to meet re-screening criteria
* Participation in a clinical research trial that included the receipt of an investigational product or any experimental therapeutic procedure within 26 weeks prior to the Screening Visit, or planned participation in any such trial
* Subjects requiring the use of opioids > 1x per week within 12 weeks prior to Day 1
* History of malignancy within the last 5 years; not including subjects with prior history of adequately treated in situ cervical cancer or basal or squamous cell skin cancer
* Clinically significant abnormal screening hematology values, blood chemistry values, or urinalysis values as determined by the Investigator
* Any known active infections, including urinary tract infection, upper respiratory tract infection, sinusitis, suspicion of IA infection, hepatitis B or hepatitis C infection, and/or infections that may compromise the immune system such as human immunodeficiency virus (HIV) at Day 1

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, M.D., Study Director — Biosplice Therapeutics, Inc.
Locations (73):
- United States (73):
  - Research Site, Birmingham, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Canoga Park, California
  - Research Site, Garden Grove, California
  - Research Site, La Mesa, California
  - Research Site, Norco, California
  - Research Site, Pomona, California
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Thousand Oaks, California
  - Research Site, Westminster, California
  - Research Site, Boulder, Colorado
  - Research Site, Hamden, Connecticut
  - Reserach Site, Clearwater, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Gulf Breeze, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Sunrise, Florida
  - Research Site, Sweetwater, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Winter Haven, Florida
  - Research Site 1, Winter Park, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Newnan, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Greenwood, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Wheaton, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Troy, Michigan
  - Research Site, Hazelwood, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site 1, St Louis, Missouri
  - Research Site 2, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Freehold, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Hartsdale, New York
  - Research Site, Rochester, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Fort Mill, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Bellaire, Texas
  - Research Site, Carrollton, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Plano, Texas
  - Research Site, Draper, Utah
  - Research Site, Ogden, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Richmond, Virginia

REFERENCES:
- [Derived] Tambiah J, Kennedy S, Swearingen C, McAlindon T, Yazici Y. Impact of structural severity on outcomes in knee osteoarthritis: an analysis of data from phase 2 and phase 3 lorecivivint clinical trials. Rheumatology (Oxford). 2025 May 1;64(5):2583-2590. doi: 10.1093/rheumatology/keae610. PMID 39495154

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle | Lorecivivint
Started | 253 | 243
Completed | 233 | 221
Not Completed | 20 | 22
Not completed — Adverse Event | 1 | 1
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 3 | 6
Not completed — Lost to Follow-up | 3 | 5
Not completed — Subject Non-Compliance | 1 | 1
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Duplicate Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | Lorecivivint | Total
Number analyzed (Participants) | 239 | 231 | 470
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (7.9) | 61.0 (8.7) | 61.0 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 136 | 284
  Male | 91 | 95 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 60 | 115
  Not Hispanic or Latino | 184 | 171 | 355
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  Black or African American | 45 | 48 | 93
  White | 181 | 167 | 348
  More than one race | 4 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0
Osteoarthritis Symptoms Laterality [Count of Participants; unit: Participants]
  Bilateral Symptoms | 170 | 149 | 319
  Unilateral Symptoms | 69 | 82 | 151
Kellgren-Lawrence Grade [Count of Participants; unit: Participants] — The Kellgren and Lawrence classification system is a common method used in research of classifying the severity of knee osteoarthritis (OA) by radiograph.
  Kellgren-Lawrence Grade has five categories, with OA deemed present at Grade 2+:
  * 0: definite absence of OA
  * 1: doubtful joint space narrowing and possible osteophytic lipping
  * 2: definite osteophytes and possible joint space narrowing
  * 3: multiple osteophytes, definite narrowing of joint space, some sclerosis
  * 4: large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity
  Participants
    Grade 2 | 115 | 111 | 226
    Grade 3 | 124 | 120 | 244
Medial Joint Space Width [Mean (Standard Deviation); unit: mm] | 2.74 (1.47) | 2.79 (1.57) | 2.77 (1.52)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline OA Pain in the Target Knee as Assessed by the Weekly Average of Daily Pain Numeric Rating Scale (NRS) at Week 12
Description: Evaluate change from baseline OA pain in the target knee as assessed by the weekly average of daily pain NRS at Week 12. The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 represents the worst possible pain.
Time Frame: Baseline and Week 12
Population: Full Analysis Set includes all subjects who were randomized and received a study injection. Subjects' observed data were analyzed as randomized without imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 213 | 211
units on a scale | -2.15 (0.14) | -2.22 (0.14)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.703, Mixed Models Analysis; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.46 to 0.31], Standard Error of Mean 0.20

2. Secondary Outcome: Change From Baseline OA Pain in the Target Knee as Assessed by the Weekly Average of Daily Pain Numeric Rating Scale (NRS) at Week 24
Description: Evaluate change from baseline OA pain in the target knee as assessed by the weekly average of daily pain NRS at Week 24. The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 represents the worst possible pain.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 201 | 185
units on a scale | -2.31 (0.14) | -2.26 (0.14)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.813, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.34 to 0.43], Standard Error of Mean 0.20

3. Secondary Outcome: Change From Baseline OA Function in the Target Knee as Assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscore (WOMAC Function) at Week 12
Description: Evaluate change from baseline OA function in the target knee as assessed by WOMAC Function subscore at Week 12. The WOMAC is a widely-used, proprietary outcome measurement tool used to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on an 11-point numeric rating scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Function raw subscore ranges from 0 to 170, and is scaled 0 (highest overall function) to 100 (lowest overall function) for analysis and reporting.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 222 | 218
units on a scale | -22.00 (1.42) | -20.29 (1.45)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.398, Mixed Models Analysis; Mean Difference (Final Values) = 1.72, 95% CI 2-sided [-2.28 to 5.71], Standard Error of Mean 2.03

4. Secondary Outcome: Change From Baseline OA Function in the Target Knee as Assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscore (WOMAC Function) at Week 24
Description: Evaluate change from baseline OA function in the target knee as assessed by WOMAC Function subscore at Week 24. The WOMAC is a widely-used, proprietary outcome measurement tool used to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on an 11-point numeric rating scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Function raw subscore ranges from 0 to 170, and is scaled 0 (highest overall function) to 100 (lowest overall function) for analysis and reporting.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 215 | 202
units on a scale | -21.91 (1.51) | -20.60 (1.55)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.544, Mixed Models Analysis; Mean Difference (Final Values) = 1.31, 95% CI 2-sided [-2.94 to 5.57], Standard Error of Mean 2.16

5. Secondary Outcome: Change From Baseline OA Disease Activity as Assessed by Patient Global Assessment at Week 12
Description: Evaluate change from baseline OA disease activity as assessed by Patient Global Assessment at Week 12. The Patient Global Assessment is an 11-point [0-10] Numeric Rating Scale [NRS] on which the subjects will rate how they feel their target knee OA is doing, considering all the ways in which their target knee OA may affect them. The NRS is anchored by descriptors at each end ("Very Good" on the left and "Very Bad" on the right). For analysis, Patient Global Assessment scores were scaled to [0-100], where 0 represents "Very Good" and 100 represents "Very Bad".
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 228 | 220
units on a scale | -22.36 (1.52) | -23.19 (1.56)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.704, Mixed Models Analysis; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-5.12 to 3.46], Standard Error of Mean 2.18

6. Secondary Outcome: Change From Baseline OA Disease Activity as Assessed by Patient Global Assessment at Week 24
Description: Evaluate change from baseline OA disease activity as assessed by Patient Global Assessment at Week 24. The Patient Global Assessment is an 11-point [0-10] Numeric Rating Scale [NRS] on which the subjects will rate how they feel their target knee OA is doing, considering all the ways in which their target knee OA may affect them. The NRS is anchored by descriptors at each end ("Very Good" on the left and "Very Bad" on the right). For analysis, Patient Global Assessment scores were scaled to [0-100], where 0 represents "Very Good" and 100 represents "Very Bad".
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 219 | 204
units on a scale | -22.18 (1.64) | -23.44 (1.69)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.594, Mixed Models Analysis; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-5.89 to 3.38], Standard Error of Mean 2.36

7. Post Hoc Outcome: Change From Baseline OA Pain in the Target Knee as Assessed by the Weekly Average of Daily Pain Numeric Rating Scale (NRS) at Week 12 in Subjects With Kellgren-Lawrence Grade 2
Description: Evaluate change from baseline OA pain in the target knee as assessed by the weekly average of daily pain NRS at Week 12 in those subjects with Kellgren-Lawrence Grade 2. The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 represents the worst possible pain.
Time Frame: Baseline and Week 12
Population: The Per-Protocol Analysis Set (PPAS) includes FAS subjects who received the correct treatment, completed the study, and did not have any protocol deviations that might impact the evaluation of efficacy outcomes. Kellgren-Lawrence Grade 2 only subjects' observed data were analyzed as randomized without imputation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 94 | 86
units on a scale | -1.77 (0.23) | -2.30 (0.24)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.115, ANCOVA; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.20 to 0.13], Standard Error of Mean 0.34

8. Post Hoc Outcome: Change From Baseline OA Pain in the Target Knee as Assessed by the Weekly Average of Daily Pain Numeric Rating Scale (NRS) at Week 24 in Subjects With Kellgren-Lawrence Grade 2
Description: Evaluate change from baseline OA pain in the target knee as assessed by the weekly average of daily pain NRS at Week 24 in those subjects with Kellgren-Lawrence Grade 2. The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 represents the worst possible pain.
Time Frame: Baseline and Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 90 | 80
units on a scale | -1.94 (0.25) | -2.60 (0.27)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.075, ANCOVA; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-1.38 to 0.07], Standard Error of Mean 0.37

9. Post Hoc Outcome: Change From Baseline OA Function in the Target Knee as Assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscore (WOMAC Function) at Week 12 in Subjects With Kellgren-Lawrence Grade 2
Description: Evaluate change from baseline OA function in the target knee as assessed by WOMAC Function subscore at Week 12 in those subjects With Kellgren-Lawrence Grade 2. The WOMAC is a widely-used, proprietary outcome measurement tool used to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on an 11-point numeric rating scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Function raw subscore ranges from 0 to 170, and is scaled 0 (highest overall function) to 100 (lowest overall function) for analysis and reporting.
Time Frame: Baseline and Week 12
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 93 | 93
units on a scale | -17.69 (2.20) | -22.94 (2.20)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.094, ANCOVA; Mean Difference (Final Values) = -5.25, 95% CI 2-sided [-11.40 to 0.90], Standard Error of Mean 3.12

10. Post Hoc Outcome: Change From Baseline OA Function in the Target Knee as Assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscore (WOMAC Function) at Week 24 in Subjects With Kellgren-Lawrence Grade 2
Description: Evaluate change from baseline OA function in the target knee as assessed by WOMAC Function subscore at Week 24 in those subjects With Kellgren-Lawrence Grade 2. The WOMAC is a widely-used, proprietary outcome measurement tool used to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on an 11-point numeric rating scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Function raw subscore ranges from 0 to 170, and is scaled 0 (highest overall function) to 100 (lowest overall function) for analysis and reporting.
Time Frame: Baseline and Week 24
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 93 | 89
units on a scale | -19.76 (2.25) | -23.60 (2.30)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.234, ANCOVA; Mean Difference (Final Values) = -3.85, 95% CI 2-sided [-10.20 to 2.51], Standard Error of Mean 3.22

11. Post Hoc Outcome: Change From Baseline OA Disease Activity as Assessed by Patient Global Assessment at Week 12 in Subjects With Kellgren-Lawrence Grade 2
Description: Evaluate change from baseline OA disease activity as assessed by Patient Global Assessment at Week 12 in those subjects with Kellgren-Lawrence Grade 2. The Patient Global Assessment is an 11-point [0-10] Numeric Rating Scale [NRS] on which the subjects will rate how they feel their target knee OA is doing, considering all the ways in which their target knee OA may affect them. The NRS is anchored by descriptors at each end ("Very Good" on the left and "Very Bad" on the right). For analysis, Patient Global Assessment scores were scaled to [0-100], where 0 represents "Very Good" and 100 represents "Very Bad".
Time Frame: Baseline and Week 12
Population: The Per-Protocol Analysis Set (PPAS) includes FAS subjects who received the correct treatment, completed the study, and did not have any protocol deviations that might impact the evaluation of efficacy outcomes. Kellgren-Lawrence Grade 2 only subjects' observed data were analyzed as randomized without imputation.)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 98 | 94
units on a scale | -17.78 (2.33) | -24.76 (2.38)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.038, ANCOVA; Mean Difference (Final Values) = -6.98, 95% CI 2-sided [-13.57 to -0.40], Standard Error of Mean 3.34

12. Post Hoc Outcome: Change From Baseline OA Disease Activity as Assessed by Patient Global Assessment at Week 24 in Subjects With Kellgren-Lawrence Grade 2
Description: Evaluate change from baseline OA disease activity as assessed by Patient Global Assessment at Week 24 in those subjects with Kellgren-Lawrence Grade 2. The Patient Global Assessment is an 11-point [0-10] Numeric Rating Scale [NRS] on which the subjects will rate how they feel their target knee OA is doing, considering all the ways in which their target knee OA may affect them. The NRS is anchored by descriptors at each end ("Very Good" on the left and "Very Bad" on the right). For analysis, Patient Global Assessment scores were scaled to [0-100], where 0 represents "Very Good" and 100 represents "Very Bad".
Time Frame: Baseline and Week 24
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Vehicle | Lorecivivint
Number analyzed (Participants) | 97 | 89
units on a scale | -18.94 (2.46) | -27.33 (2.56)
Statistical Analysis 1: Comparison: Vehicle vs Lorecivivint; Test type: Superiority; p = 0.019, ANCOVA; Mean Difference (Final Values) = -8.39, 95% CI 2-sided [-15.40 to -1.38], Standard Error of Mean 3.55

ADVERSE EVENTS:
Time Frame: AEs were assessed at each clinic visit from the time of study medication injection on Day 1 through Week 28 (EOS) or Early Termination.
Arm/Group | Vehicle | Lorecivivint
All-Cause Mortality (participants affected / at risk) | 1/251 | 0/241
Serious Adverse Events (participants affected / at risk) | 1/251 | 4/241
Other Adverse Events (participants affected / at risk) | 38/251 | 27/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=251) | Lorecivivint (N=241)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=251) | Lorecivivint (N=241)
Urinary tract infection (Infections and infestations) | 7 (9) | 9 (13)
COVID-19 (Infections and infestations) | 8 (8) | 7 (8)
Hypertension (Vascular disorders) | 3 (3) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (16) | 7 (7)
Headache (Nervous system disorders) | 5 (6) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
This trial was conducted during COVID-19 and its confounding effects on clinical outcomes in knee OA patients based on observational data have been reported (Knee Surg Sports Traumatol Arthrosc, 2020;28(8):2435-43). Structural progression enrichment in the OA-11 trial, which enrolled concurrently, might have confounded short-term therapeutic pain detection; this hypothesis was evaluated in the post-hoc Kellgren-Lawrence Grade 2 only analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT04385303/Prot_001.pdf
  • Statistical Analysis Plan (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT04385303/SAP_002.pdf